CLINICAL TRIAL: NCT00004980
Title: Repetitive Transcranial Magnetic Stimulation of Speech Processing Brain Areas in Schizophrenic Patients Who Hear "Voices"
Brief Title: Repetitive Transcranial Magnetic Stimulation for "Voices"
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R21MH063326 (NIH); R21MH063326 (NIH); YALESM-9281; 199/14809; A5-ETPD
Record Dates: First submitted 2000-03-10; First posted 2000-03-13 (Estimated); Results first posted 2012-07-09 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Schizophrenia
Keywords: neurologic and psychiatric disorders; rare disease; schizophrenia
MeSH Terms: conditions — Schizophrenia; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active rTMS (Experimental): 1-Hz rTMS delivered to left temporoparietal cortex at 90% motor threshold for 16 minutes per session given one session per day for nine consecutive days (with the exception of weekends)
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- sham stimulation (Placebo Comparator): Sham stimulation delivered 16 minutes per session given one session per day for nine consecutive days (with the exception of weekends)
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) — a total of 132 minutes of stimulation at one hertz, motor threshold set at 80%, delivered to TP3 scalp site
  Other Names: MATSTIM SUPER RAPID
  Arms: active rTMS
Device: sham stimulation — 132 minutes of stimulation given at 80% motor threshold with coil tilted "single wing" 45 degrees away from scalp deliverd to TP3 site
  Other Names: MAGSTIM SUPER RAPID
  Arms: sham stimulation

SUMMARY:
OBJECTIVES:

I. Determine the effect of repetitive transcranial magnetic stimulation on treatment refractory auditory hallucinations of patients with schizophrenia.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind study. Patients are randomized to one of two treatment arms.

Group I: Patients receive 9 sessions of active transcranial magnetic stimulation (rTMS) which consists of 8 minutes of rTMS during session 1, 12 minutes duration during session 2, and 16 minutes duration during sessions 3-9. The total duration of stimulation is 132 minutes. Each session was given on a separate day and in general each session occurred on consecutive days with the exception of weekends.

Group II: Patients receive 9 sessions of sham stimulation, which consists of 8 minutes of sham stimulation during session 1, 12 minutes duration sham stimulation during session 2, and 16 minutes duration sham stimulation during sessions 3-9. The total duration of sham stimulation is 132 minutes. Each session was given conducted on a separate day and in general each session occured on consecutive days with the exception of weekends.

This study provided pilot data supplying the basis for our current study - NCT00308997 -- see our website for details

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Inclusion criteria:

* Diagnosis of schizophrenia or schizoaffective disorder based on DSM-IV version of SCID
* Auditory hallucinations of spoken speech occurring at least 5 times per day where subject able to discern verbal content
* Right-handed
* At least 4 weeks on stable antipsychotic medication

Exclusion criteria:

* history of seizure (unless due to drug withdrawal or medication that is no longer prescribed)
* history of epilepsy in first degree relatives
* estimated IQ less than 80
* unable to provide informed consent
* significant unstable medical condition
* current treatment with clozapine or bupropion
* cochlear implants or other metal in the head (surgical, etc.)
* history of cardiac arrhythmia
* cardiac pacemaker
* active drug or alcohol abuse within prior 6 weeks
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 1999-12; Primary Completion 2005-01 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Hoffman, Study Chair — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Result] Hoffman RE, Gueorguieva R, Hawkins KA, Varanko M, Boutros NN, Wu YT, Carroll K, Krystal JH. Temporoparietal transcranial magnetic stimulation for auditory hallucinations: safety, efficacy and moderators in a fifty patient sample. Biol Psychiatry. 2005 Jul 15;58(2):97-104. doi: 10.1016/j.biopsych.2005.03.041. PMID 15936729
- See also: Click here for the Yale School of Medicine Web site describing current, on-going rTMS trial for auditory hallucinations — http://psychiatry.yale.edu/research/programs/clinical_people/rtms.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Repetitive Transcanial Magnetic Stimulation: Participants received active repetitive transcranial magnetic stimulation (rTMS)
- Placebo: Participants received sham stimulation
Period: Overall Study
Arm/Group | Active Repetitive Transcanial Magnetic Stimulation | Placebo
Started | 27 | 23
Completed | 25 | 21
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — memory difficulties | 1 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Repetitive Transcanial Magnetic Stimulation | Placebo | Total
Number analyzed (Participants) | 27 | 23 | 50
Age Continuous [Mean (Standard Deviation); unit: Years] | 35.1 (11.9) | 35.5 (9.5) | 35.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 18 | 15 | 33
Medication Resistance [Number; unit: Participants] — Number of participants who were medication resistant
  Participants
    Medication Resistant | 21 | 18 | 39
    Not Medication Resistant | 6 | 5 | 11
Total Auditory Hallucination Rate Scale (AHRS) score [Mean (Standard Deviation); unit: Scores on a scale] — Sum of 7 variables: frequency of hallucinations, reality of hallucinations, loudness of hallucinations, number of acoustically distinct voices, length of hallucinations, attentional salience of hallucinations, level of distress induced by hallucinations; higher score connotes more severe hallucinations; lowest score is 4, highest score is 37
  Scores on a scale | 25.1 (5.0) | 26.1 (5.7) | 25.6 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Hallucination Change Score (HCS) After 9 Active/Sham rTMS Sessions
Description: Change in hallucination severity relative to baseline with scores ranging 1 in unit intervals to 20 anchored as follows: 0=hallucinations stopped, 10=no change, 20=hallucinations twice as severe as baseline
Time Frame: After the 9th active/sham rTMS session (up to 2 weeks or end of intervention)
Population: Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Active Repetitive Transcanial Magnetic Stimulation | Placebo
Number analyzed (Participants) | 27 | 23
Units on a scale | 5.85 (2.85) | 8.61 (3.80)
Statistical Analysis 1: Comparison: Active Repetitive Transcanial Magnetic Stimulation vs Placebo; Test type: Superiority or Other; p = .005, t-test, 2 sided — a priori threshold for statistical significance was .05; degree of freedom = 48; Mean Difference (Final Values) = -2.76, 95% CI [-4.65 to -.86], Standard Error of Mean .514

2. Secondary Outcome: Change From Baseline in Hallucination Frequency After 9 Active/Shame rTMS Sessions
Description: Difference between baseline hallucination frequency and hallucintion frequency at last assessment. Assessed on the basis of a 0-9 scale, with higher scores being more severe.
Time Frame: After the 9th active/sham rTMS session (up to 2 weeks or end of intervention)
Population: LOCF
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Active Repetitive Transcanial Magnetic Stimulation | Placebo
Number analyzed (Participants) | 27 | 23
Score on a scale | 1.42 (1.49) | .15 (1.14)
Statistical Analysis 1: Comparison: Active Repetitive Transcanial Magnetic Stimulation vs Placebo; null hypothesis is that the groups are the same; Test type: Superiority or Other; p = .002, t-test, 2 sided — a priori threshold for statistical significance was .05; degrees of freedom = 48; Mean Difference (Final Values) = 1.27, 95% CI [.507 to 2.03], Standard Error of Mean .327

3. Secondary Outcome: Clinical Global Improvement (CGI) Scale After 9 Active/Shame rTMS Sessions
Description: Scaled from 1-7 as follows: 1=dramatically improved, 2=moderately improved, 3=minimally improved, 4=no change, 5=minimally worsened, 6=moderately worsened, 7=dramatically worsened
Time Frame: After the 9th active/sham rTMS session (up to 2 weeks or end of intervention)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Active Repetitive Transcanial Magnetic Stimulation | Placebo
Number analyzed (Participants) | 26 | 22
Units on a scale | 2.84 (.845) | 3.79 (.882)
Statistical Analysis 1: Comparison: Active Repetitive Transcanial Magnetic Stimulation vs Placebo; Test type: Superiority or Other; p = .001, t-test, 2 sided — A priori threshold for statistical significance was .05; degrees of freedom = 46; Median Difference (Final Values) = -.949, 95% CI [-1.45 to -.44], Standard Error of Mean .524

4. Secondary Outcome: Responder Status
Description: Responder defined as a participant who attains an endpoint hallucination change score (HCS) of 5 or lower after 9 active/shame rTMS sessions.
  Change in hallucination severity relative to baseline with scores ranging 1 in unit intervals to 20 anchored as follows: 0=hallucinations stopped, 10=no change, 20=hallucinations twice as severe as baseline
Time Frame: After the 9th active/sham rTMS session (up to 2 weeks or end of intervention)
Population: LOCF
Measure: Number; unit: Participants
Arm/Group | Active Repetitive Transcanial Magnetic Stimulation | Placebo
Number analyzed (Participants) | 27 | 23
Participants | 14 | 4
Statistical Analysis 1: Comparison: Active Repetitive Transcanial Magnetic Stimulation vs Placebo; Test type: Superiority or Other; p = .01, Chi-squared — a priori threshold for statistical significance = .05

ADVERSE EVENTS:
Time Frame: Adverse event reporting was collected for the duration of the study (41 months)
Description: Adverse events were systematically collected with focused questions each day during the trial
Arm/Group | Active Repetitive Transcanial Magnetic Stimulation | Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/23
Other Adverse Events (participants affected / at risk) | 16/27 | 3/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Repetitive Transcanial Magnetic Stimulation (N=27) | Placebo (N=23)
Headache (Nervous system disorders) | 16 | 3 — Transient headache and responsive to acetaminophen

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No